CLINICAL TRIAL: NCT03478202
Title: An Open-Label Pilot Study Evaluating the Effect of the GOLO for Life Weight Management Program on Weight and Metabolic Syndrome Indicators in Patients With Type II Diabetes Mellitus
Brief Title: GOLO Open-Label Pilot 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Golo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GOLO1701
Record Dates: First submitted 2018-03-19; First posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Label RELEASE Supplement (Experimental)
  Interventions: Dietary Supplement: GOLO RELEASE

INTERVENTIONS:
Dietary Supplement: GOLO RELEASE — GOLO RELEASE plus Diet

SUMMARY:
The objective of this open-label pilot study is to evaluate the effect of the commercially available GOLO for Life (GFL) weight management program on body weight in a type 2 diabetic patient population after approximately 3 months.

DETAILED DESCRIPTION:
Golo For Life (GFL) is a weight management program that helps people who are overweight or obese limit and portion their consumption of conventional foods and make healthier choices in their diets. GFL includes a point-based system from the four macronutrient food groups that is based on the individual's activity level and body mass. Additionally, GFL includes common-sense instructions, motivation and tips supporting compliance and requires a minimum of 15 minutes of exercise per day. GFL also includes a dietary supplement containing zinc and chromium, essential nutrients that support regulation of blood sugar.

In case studies from clinician and wellness program use, GFL has shown the ability to reduce body weight in both healthy and diabetic people who are overweight or obese. Secondary endpoints including measures of blood sugar have been observed to decrease as a result of the GFL program.

While GFL has been developed and used in private clinical practice in both healthy overweight and type 2 diabetic people, more systematic research is needed to determine to what extent it is able to support healthy weight loss. This open-label pilot study is intended to observe the effects of the program in a representative group of subjects with stable type 2 diabetes at one outpatient medical practice.

The objective of this open-label pilot study is to evaluate the effect of the commercially available GOLO for Life (GFL) weight management program on body weight in a type 2 diabetic patient population after approximately 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 69 years
* Diagnosis of type 2 diabetes mellitus at least six months prior to enrollment
* Currently being treated for type 2 diabetes mellitus with oral medication or diet therapy
* Oral medications or diet therapy for diabetes stable for at least three months prior to enrollment
* Body mass index (BMI) ≥ 30 and ≤ 45 kg/m2
* Have the ability to engage in at least 15 minutes of moderate physical activity such as brisk walking
* Willing to comply with study procedures described herein

Exclusion Criteria:

* Current uncontrolled type 2 diabetes (clinically significant increases in FBG or HbA1c in the past 6 months, as determined by a physician or other appropriate clinical measure)
* Subjects with a history of hypoglycemia
* A history of an eating disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* Known allergy to any of the components in the GOLO for Life supplement
* A history of prior surgery for weight loss
* Currently taking injectable medications to control diabetes, including insulin and GLP-1 agonists
* Current diagnosis with Type 1 diabetes mellitus
* Currently pregnant or breastfeeding or have had a baby within the last six weeks
* Planning to become pregnant in the next three months. Women of child bearing potential must be willing and able to use adequate and reliable contraception throughout the study (e.g. abstinence or barrier with additional spermicidal foam or jelly, or the use of intrauterine device or hormonal contraception).
* Clinically unstable heart disease or uncontrolled hypertension at screening defined as Systolic blood pressure greater than 180 mmHG or Diastolic blood pressure greater than 100 mmHG
* Current clinical diagnosis of unstable or uncontrolled kidney or liver disease, cancer, chronic neurological disease.
* Current participation in any other weight loss or weight management program
* Currently taking weight loss medications, or medications or supplements known to be associated with significant weight loss or weight gain
* Has any condition that, in the opinion of the investigator, would make participation in this study not in the best interest of the subject or that could prevent, limit or confound the protocol-specified assessments. Examples include: history of diabetic ketoacidosis; active chronic liver disease or cirrhosis; chronic autoimmune disease; inflammatory bowel disease, colonic ulceration, partial intestinal obstruction, subjects predisposed to intestinal obstruction; chronic intestinal diseases associated with marked disorders of digestion or absorption

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-12-23 (Actual); Study Completion 2017-12-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline in weight | 3 months

SECONDARY OUTCOMES:
Change from baseline in waist circumference | 3 months
Change from baseline in hip circumference | 3 months
Change from baseline in Body Mass Index (BMI) | 3 months
Change from baseline in Hemoglobin A1C | 3 months
Change from baseline in fasting Insulin level | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Buynak Clinical Research, Valparaiso, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided